CLINICAL TRIAL: NCT01198132
Title: A Multicentre, Randomised, Double-blind, Placebo-controlled Study of the Efficacy of Supplementary Treatment With Cholecalciferol (Vitamin D3) in Patients With Relapsing- Multiple Sclerosis (RMS) Treated With Subcutaneous Interferon Beta-1a 44 µg 3 Times Weekly
Brief Title: A Multicentre Study of the Efficacy and Safety of Supplementary Treatment With Cholecalciferol in Patients With Relapsing Multiple Sclerosis Treated With Subcutaneous Interferon Beta-1a 44 µg 3 Times Weekly
Acronym: CHOLINE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck Serono S.A.S, France (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 701068-524; 2009-013695-46 (EudraCT Number)
Record Dates: First submitted 2010-09-08; First posted 2010-09-09 (Estimated); Results first posted 2017-12-14 (Actual); Last update posted 2017-12-14 (Actual); Status verified 2017-05

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis Relapsing-Remitting; Relapsing Multiple Sclerosis (RMS); Rebif; Vitamin D3; Cholecalciferol
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting | interventions — Cholecalciferol; Interferon beta-1a

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cholecalciferol (Experimental): Subjects receive Cholecalciferol 100,000 IU one dose fortnightly (equivalent to a daily dose of approximately 7142 IU) for 96 weeks treatment period along with subcutaneous Rebif 3 times a week.
  Interventions: Dietary Supplement: Cholecalciferol (Vitamin D3); Drug: Rebif
- Placebo (Placebo Comparator): Subjects receive matching placebo to Cholecalciferol once every two weeks along with subcutaneous injection of Rebif 3 times weekly.
  Interventions: Dietary Supplement: Placebo; Drug: Rebif

INTERVENTIONS:
Dietary Supplement: Cholecalciferol (Vitamin D3) — Subjects receive Cholecalciferol 100,000 IU one dose fortnightly (equivalent to a daily dose of approximately 7142 IU) for 96 weeks treatment period along with subcutaneous Rebif 44 mcg 3 times a week.
  Other Names: Vitamin D3
  Arms: Cholecalciferol
Dietary Supplement: Placebo — Subjects receive matching placebo to Cholecalciferol once every two weeks orally along with subcutaneous injection of Rebif 44 mcg 3 times weekly.
  Arms: Placebo
Drug: Rebif — Subjects receive subcutaneous injection of Rebif 44 mcg 3 times weekly.
  Other Names: Interferon beta-1a

SUMMARY:
The aim of this multicentre, randomised, double-blind, placebo-controlled study is to evaluate the efficacy and safety of supplementary treatment with cholecalciferol (vitamin D3) in subjects with relapsing multiple sclerosis (R MS) treated with subcutaneous (s.c.) interferon beta-1a 44 microgram (mcg) [Rebif] 3 times weekly. The subjects will be divided into 2 groups, one receiving cholecalciferol 100,000 IU twice monthly along with Rebif treatment and the other group will be on placebo along with Rebif treatment. A total of 200 subjects will be recruited in 20-30 centres in France.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of RRMS according to Poser criteria (clinically definite multiple sclerosis [CDMS] or laboratory supported definite multiple sclerosis [LSDMS]) or according to McDonald criteria (2005).
* Subjects aged between 18 and 65 years.
* Treated with interferon beta-1a 44 mcg (or 22 mcg in case of intolerance to 44 mcg) 3 times weekly subcutaneously for 4 months ± (2 months) at the randomization visit (V1).
* Expanded disability status scale (EDSS) score between 0 and 5.
* At least one documented episode during the last two year.
* Stable disease with no episodes over the last 30 days.
* Serum 25-hydroxyvitamin D less than (<) 75 nanomolar per liter (nmol/l) at randomization visit.
* Women must not be pregnant or breast-feeding, and women of childbearing age must meet the following criteria:

  * Surgically sterilised, or
  * Using a highly effective contraceptive method throughout the entire duration of the study. A highly effective contraceptive method is defined as a method with a very low failure rate (i.e. < 1 % per year) with regular and appropriate use, e.g. implants, injectable contraceptives, combined oral contraceptives, coil, abstinence or vasectomised partner.
  * Menopausal women may be included.
* Affiliated to French healthcare insurance.
* Subjects must be ready and able to provide informed consent and comply with the protocol requirements.

Exclusion Criteria:

* Hormonal abnormalities associated with vitamin D other than low dietary intake or reduced exposure to sun, for example malabsorption (coeliac disease, Whipple's disease, inflammatory bowel disease, intestinal derivation, short bowel syndrome), cirrhosis, nephrotic syndrome, hyperthyroidism, rickets, hypoparathyroidism, cancer, granulomatous diseases (sarcoidosis, silicosis) and lymphomas known at the initial visit.
* Patients with osteoporosis or known osteopenia.
* Use of medicines affecting vitamin D metabolism other than corticosteroids, e.g. anticonvulsants (phenobarbital, primidone, phenytoin), rifampicin, isoniazid, ketoconazole, 5-FU and leucovorin, or thiazide diuretics.
* Previous or ongoing hypercalcaemia.
* Situations involving increased susceptibility to hypercalcaemia, e.g. known cardiac arrhythmia or cardiac disease, treatment with digitalis, renal lithiasis.
* Any contraindication to the treatment (cholecalciferol) stated in the summary of product characteristics.
* Moderate renal impairment defined as creatinine clearance between 30 and 60 ml/min.
* An active episode during the month prior to inclusion in the study.
* Inadequate liver function, defined as total bilirubin, aspartate aminotransferase (AST), alanine aminotransferase (ALT) or alkaline phosphatase greater than (>) 2.5 * upper limit of normal.
* Severe renal impairment defined as creatinine clearance below 30 milliliter per minute (ml/min).
* Inadequate marrow reserves, defined as white blood cells < 0.5 * lower limit of normal.
* Serious or acute heart disease such as uncontrolled cardiac arrhythmia, uncontrolled angina, cardiomyopathy or uncontrolled congestive heart failure.
* History of severe depression, or attempted suicide or ongoing suicidal ideation.
* Epilepsy inadequately controlled by treatment.
* Ongoing or previous alcohol or drug abuse (within the last two years).
* Major medical or psychiatric disease which, in the opinion of investigator, would place the subject at risk or could adversely affect compliance with the study protocol.
* Known hypersensitivity to gadolinium and/or known inability to undergo MRI.
* Any medical condition requiring chronic treatment with systemic corticosteroids.
* Participation in any other studies involving other study products over the 30 days prior to inclusion in this study.
* Legal incapacity or limited legal capacity.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2009-11 (Actual); Primary Completion 2015-03 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck KGaA, Darmstadt, Germany
Locations (1):
- CHU Hôpital Gui de Chauliac Service de Neurologie B, Montpellier, France

REFERENCES:
- [Derived] Camu W, Lehert P, Pierrot-Deseilligny C, Hautecoeur P, Besserve A, Jean Deleglise AS, Payet M, Thouvenot E, Souberbielle JC. Cholecalciferol in relapsing-remitting MS: A randomized clinical trial (CHOLINE). Neurol Neuroimmunol Neuroinflamm. 2019 Aug 6;6(5):e597. doi: 10.1212/NXI.0000000000000597. Print 2019 Sep. PMID 31454777

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 129 subjects were randomized. Out of which 126 subjects treated in the study and 90 subjects completed the study.
Groups:
- Cholecalciferol: Subjects received Cholecalciferol 100,000 IU one dose fortnightly (equivalent to a daily dose of approximately 7142 IU) for 96 weeks treatment period along with subcutaneous Rebif 44 mcg 3 times a week.
- Placebo: Subjects received matching placebo to Cholecalciferol once every two weeks orally along with subcutaneous injection of Rebif 44 mcg 3 times weekly.
Period: Overall Study
Arm/Group | Cholecalciferol | Placebo
Started | 63 | 66
Completed | 45 | 45
Not Completed | 18 | 21
Not completed — Withdrawal by Subject | 4 | 5
Not completed — Physician Decision | 5 | 4
Not completed — Other Unspecified | 3 | 6
Not completed — Lack of Efficacy | 2 | 3
Not completed — Sign/symptoms of underlying disease | 2 | 1
Not completed — Abnormal/clinically significant biologic | 1 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) set included all randomized subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cholecalciferol | Placebo | Total
Number analyzed (Participants) | 63 | 66 | 129
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.5 (9.29) | 36.9 (8.34) | 37.7 (8.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 39 | 89
  Male | 13 | 27 | 40

OUTCOME MEASURES:

1. Primary Outcome: Annualized Relapse Rate
Description: The annualized relapse rate was calculated for each treatment group as follows: the number of relapses observed during the study period divided by the time spent in the study (in years).
Time Frame: 2 years post treatment (IMP) administration
Population: ITT set included all randomized subjects.
Measure: Mean (95% Confidence Interval); unit: Relapse per year
Arm/Group | Cholecalciferol | Placebo
Number analyzed (Participants) | 63 | 66
Relapse per year | 0.45 [0.20 to 0.69] | 0.34 [0.22 to 0.46]
Statistical Analysis 1: Comparison: Cholecalciferol vs Placebo; Test type: Superiority or Other; p = 0.3797, Poisson log-linear model; Rate ratio = 0.80, 95% CI 2-sided [0.48 to 1.32]

2. Secondary Outcome: Time to First Documented Relapse
Description: Time to First Documented Relapse was calculated using Kaplan-Meier survival methods.
Time Frame: 2 years post treatment (IMP) administration
Population: ITT set included all randomized subjects. Here "Number of participant analyzed" signifies those subjects who were evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: weeks
Groups:
- Rebif +Placebo: Subjects received matching placebo to Cholecalciferol once every two weeks orally along with subcutaneous injection of Rebif 44 mcg 3 times weekly.
Arm/Group | Cholecalciferol | Rebif +Placebo
Number analyzed (Participants) | 61 | 65
weeks | NA [NA to NA] — Median and Confidence interval could not be calculated due to a limited number of events . | NA [60.1 to NA] — Median and Confidence interval could not be calculated due to a limited number of events .

3. Secondary Outcome: Mean Number of Relapses Per Subject
Description: Relapse was defined as new, worsening or recurrent neurological symptoms attributed to multiple sclerosis that last for at least 24 hours without fever or infection, or adverse reaction to prescribed medication, preceded by a stable or improving neurological status of at least 30 days. Mean and standard deviation were reported.
Time Frame: 2 years post treatment (IMP) administration
Population: ITT set included all randomized subjects.
Measure: Mean (Standard Deviation); unit: relapses
Arm/Group | Cholecalciferol | Placebo
Number analyzed (Participants) | 63 | 66
relapses | 0.5 (0.78) | 0.5 (0.75)

4. Secondary Outcome: Number of Relapse-Free (Documented) Subjects
Description: The relapse-free patients after 2 years of treatment was calculated using Cochran-Mantel-Haenszel test using the site as control variable.
Time Frame: 2 years post treatment (IMP) administration
Population: ITT set included all randomized subjects. Here "Number of participants analyzed" signifies those subjects who were evaluable for this outcome measure.
Measure: Number; unit: subjects
Arm/Group | Cholecalciferol | Placebo
Number analyzed (Participants) | 45 | 46
subjects | 35 | 27

5. Secondary Outcome: Cumulative Probability of Progression of Disability (Kaplan-Meier Curves)
Description: Disability progression was assessed using Expanded disability status scale (EDSS). EDSS assesses disability in 8 functional systems. An overall score ranging from 0 (normal) to 10 (death due to MS) was calculated. A one-point increase on the EDSS scale was considered as a progression in disability. The time to disability progression was summarized using Kaplan-Meier survival methods. The cumulative probability of confirmed disease progression at each visit was obtained by applying a Kaplan-Meier method to the time to confirmed disease progression.
Time Frame: Baseline up to week 96
Population: as for outcome 2
Measure: Number; unit: percentage of subjects
Arm/Group | Cholecalciferol | Placebo
Number analyzed (Participants) | 60 | 65
percentage of subjects | 12.7 | 9.1

6. Secondary Outcome: Number of New or Extended Lesions by T1- and T2-Weighted Magnetic Resonance Imaging (MRI)
Time Frame: 2 years post treatment (IMP) administration
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | Cholecalciferol | Placebo
Number analyzed (Participants) | 44 | 41
lesions
  T1-weighted MRI | 0.4 (0.76) | 1.9 (3.76)
  T2-weighted MRI | 0.5 (0.79) | 2.0 (4.71)

7. Secondary Outcome: Changes From Baseline in Measured Lesion Load (T2)
Description: Baseline defined as last value recorded prior to first intake of study drug.
Time Frame: Baseline, Week 96
Population: ITT set included all randomized subjects. Here "n" signifies those subjects who were evaluable for this outcome measure at the specified time points.
Measure: Mean (Standard Deviation); unit: cubic millimeter (mm^3)
Arm/Group | Cholecalciferol | Placebo
Number analyzed (Participants) | 63 | 66
cubic millimeter (mm^3)
  Baseline (n=49, 43) | 5305.4 (10858.86) | 3520.1 (4954.44)
  Change at Week 96 (n=44, 38) | -315.0 (2523.97) | 596.3 (2034.80)

8. Secondary Outcome: Change From Baseline in Measurement and Evaluation of Cognitive Ability by Paced Auditory Serial Addition Task (PASAT) Total Score At Week 96
Description: The Adapted Paced Auditory Serial Addition Task (PASAT) is a measure of cognitive function that specifically assesses auditory information processing speed and flexibility, as well as calculation ability. The total score for PASAT is the total number of correct answers (out of 60, for a total possible score ranging from 0-60 with higher score indicates higher auditory processing speed) for each trial. Change from baseline in PASAT total score at Week 96 was summarized.
Time Frame: Baseline, Week 96
Population: ITT set included all randomized subjects.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo: Subjects received matching placebo to Cholecalciferol once every two weeks orally along with sub-cutaneous injection of Rebif 44 mcg 3 times weekly.
Arm/Group | Cholecalciferol | Placebo
Number analyzed (Participants) | 63 | 66
units on a scale
  Baseline | 39.9 (14.80) | 43.3 (12.49)
  Change at Week 96 | 6.4 (8.49) | 6.0 (8.02)

9. Secondary Outcome: Change From Baseline in Euro Quality of Life Scale (EuroQol) 5-Dimension-3 Level (EQ-5D-3L)
Description: The EQ-5D health questionnaire is a generic self-reported health-related quality of life instrument that includes a 100 mm Visual Analog Scale (VAS) to measure the general health state, as well as 5 items corresponding to one dimension each: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. In this study, the VAS scale is not collected and the version 3L of the scale was used: Each dimension had 3 possible levels: 1 = no problem, 2 = some problems and 3 = extreme problems. EQ-5D-3L weighted health state index exists that combines the score of the 5 dimensions and ranges from 0 to 1 (full health). The variables for the 5 dimensions of the EQ-5D descriptive system was named 'mobility','selfcare', 'activity', 'pain', and 'anxiety'. The 5 variables contained the values for the different dimensions in the EQ-5D health profile (i.e. 1, 2, or 3).
Time Frame: 2 years post treatment (IMP) administration
Population: ITT set included all randomized subjects.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cholecalciferol | Placebo
Number analyzed (Participants) | 63 | 66
units on a scale
  Baseline (n=60, 63) | 0.7834 (0.24090) | 0.7937 (0.21447)
  Change at Week 96 (n=43, 45) | -0.0051 (0.13742) | 0.0043 (0.19654)

10. Secondary Outcome: Number of Subjects With Treatment Emergent Adverse Events (TEAEs), Serious TEAEs and Abnormal Clinical Laboratory
Description: A serious TEAE was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect and TEAE was defined as newly occurring or worsening after first dose. Clinical laboratory abnormalities are expected to be reported as adverse events if they met any criterion for seriousness, led to treatment discontinuation, required a medical intervention or were considered clinically significant by the investigator.
Time Frame: Baseline up to end of treatment (week 96)
Population: Safety set included all subjects who receive at least one administration of trial medication.
Measure: Number; unit: subjects
Arm/Group | Cholecalciferol | Placebo
Number analyzed (Participants) | 61 | 65
subjects
  TEAEs | 43 | 35
  Serious TEAEs | 11 | 10

ADVERSE EVENTS:
Time Frame: Baseline till the end of the study (week 96)
Description: Adverse events were collected for Safety population. Safety set included all subjects who receive at least one administration of trial medication.
Arm/Group | Cholecalciferol | Placebo
Serious Adverse Events (participants affected / at risk) | 11/61 | 10/65
Other Adverse Events (participants affected / at risk) | 40/61 | 31/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cholecalciferol (N=61) | Placebo (N=65)
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Stress cardiomyopathy (Cardiac disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Abdominal abscess (Infections and infestations) | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Epilepsy (Nervous system disorders) | 1 | 0
Pregnancy on contraceptive (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Pregnancy on oral contraceptive (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Pregnancy after post coital contraception (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Foetal death (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Abortion induced complete (Surgical and medical procedures) | 1 | 0
Plastic surgery to the face (Surgical and medical procedures) | 1 | 0
Adrenal mass (Endocrine disorders) | 0 | 1
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cholecalciferol (N=61) | Placebo (N=65)
Urinary tract infection (Infections and infestations) | 4 | 4
Nasopharyngitis (Infections and infestations) | 3 | 4
Bronchitis (Infections and infestations) | 1 | 4
Gastroenteritis (Infections and infestations) | 1 | 4
Headache (Nervous system disorders) | 4 | 1
Influenza like illness (General disorders) | 1 | 5
Asthenia (General disorders) | 4 | 2
Depression (Psychiatric disorders) | 5 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Influenza (Infections and infestations) | 3 | 1
Cystitis (Infections and infestations) | 2 | 0
Gingivitis (Infections and infestations) | 2 | 0
Hordeolum (Infections and infestations) | 1 | 0
Oral candidiasis (Infections and infestations) | 1 | 0
Oral herpes (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 2
Paronychia (Infections and infestations) | 1 | 0
Tooth abscess (Infections and infestations) | 1 | 0
Tooth infection (Infections and infestations) | 1 | 0
Tracheobronchitis (Infections and infestations) | 1 | 0
Bronchitis viral (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1
Migraine (Nervous system disorders) | 3 | 1
Dizziness (Nervous system disorders) | 1 | 0
Optic neuritis (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 1
Radiculitis (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 0 | 1
Injection site erythema (General disorders) | 2 | 0
Injection site pain (General disorders) | 1 | 0
Injection site reaction (General disorders) | 1 | 2
Malaise (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Cyst (General disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Articular calcification (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 2 | 0
Depressive symptom (Psychiatric disorders) | 0 | 1
Stress (Psychiatric disorders) | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 2 | 0
Transaminases increased (Investigations) | 2 | 0
Creatinine urine increased (Investigations) | 1 | 0
Serum ferritin increased (Investigations) | 1 | 0
Urine calcium/creatinine ratio increased (Investigations) | 1 | 0
White blood cell count decreased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 0 | 1
Creatinine renal clearance decreased (Investigations) | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 1
Normetanephrine urine increased (Investigations) | 0 | 1
Weight increased (Investigations) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Aphthous stomatitis (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Gingival pain (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 2
Dental discomfort (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 3 | 0
Head injury (Injury, poisoning and procedural complications) | 2 | 0
Breast injury (Injury, poisoning and procedural complications) | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 2
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 1
Spinal column injury (Injury, poisoning and procedural complications) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Snoring (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Skin necrosis (Skin and subcutaneous tissue disorders) | 2 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Skin reaction (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Menopause (Social circumstances) | 3 | 0
Dyslipidaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Metabolic syndrome (Metabolism and nutrition disorders) | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 1 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1
Diabetes insipidus (Endocrine disorders) | 1 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Hypertension (Vascular disorders) | 1 | 1
Arterial disorder (Vascular disorders) | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1
Eye pain (Eye disorders) | 0 | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first publication will be publication of results of the analysis of primary endpoint(s) that will include data from all trial centers. Any publications and presentations of results, either in whole or in part, by investigators or their representatives will require pre-submission review by the sponsor/CRO. Sponsor will not suppress or veto publications, but maintains right to delay publication in order to protect intellectual property rights.